CLINICAL TRIAL: NCT03082664
Title: Topical Negative Pressure Wound Therapy to Prevent Wound Complications Following Cesarean Section in High Risk Obstetric Patients
Brief Title: Negative Pressure Wound Therapy to Prevent Wound Complications Following Cesarean Section in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Meghan Hill, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1412596588
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: High Risk Pregnancy; Cesarean Wound Disruption With Postnatal Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard dressing (No Intervention): Standard dressing will be applied after C-section.
- PICO dressing (Experimental): Device: PICO Single Use Negative Pressure Wound Therapy
  Interventions: Device: PICO Single Use Negative Pressure Wound Therapy

INTERVENTIONS:
Device: PICO Single Use Negative Pressure Wound Therapy — The PICO device will be placed over the closed cesarean section incision.
  Other Names: Smith & Nephew PICO patch
  Arms: PICO dressing

SUMMARY:
This is a randomized controlled trial. Patients with a condition that increases their risk of a wound complication will be approached for inclusion in the trial. Each participant agreeing to study inclusion will be randomized to either suture alone or to closure of their skin incision with suture and then with prophylactic placement of a wound vac (PICO).

DETAILED DESCRIPTION:
Once consent has been obtained from patients, an envelope containing the study allocation will be retrieved from the Pyxis.

* Non-wound vac patients will undergo wound closure with subcutaneous fat closure with Vicryl in all cases that this is practicable (in extremely thin patients, this may not be possible), followed by subcuticular skin closure also using Vicryl. A compression dressing will then be applied. This dressing is usually removed by the clinician the following day.
* Wound vac (PICO) patients will undergo wound closure with subcutaneous fat closure with Vicryl in all cases that this is practicable (in extremely thin patients, this may not be possible), followed by subcuticular skin closure also using Vicryl. The wound vac system will then be applied over the closed incision. This vac dressing will then be removed on the day of hospital discharge and replaced with a second bandage and the wound vacuum will be re-activated. The patient will remove the bandage and discard on POD#7. This is per the manufacturer's guidelines for length of use.
* If the patient fails the wound vac therapy- ie the wound separates and requires traditional wound care (packing, wet to dry dressing, etc), then the PICO system is no longer used as part of their care.

It would be unrealistic to try to standardize the entire operative approach (closure of the uterus, closure of the fascia) as the different providers working at the hospital may choose not to participate if the approach specified deviated too much from their usual technique. Different providers may typically use different kinds or sutures (made of different material, and of different sizes) or staples to close the subcutaneous fat and the skin. However, for this study all patients will have the subcutaneous fat and skin closed in the same manner (with Vicryl suture). To participate in the trial patients will have to agree to these closure materials. For this study a standard closure with suture was chosen as there is evidence suggesting a lower rate of wound complications with suture as compared to staples.

The wound will be re-assessed at their 2 week and 6 week post-op follow up visits. The patients will be assessed by a physician at their post-operative clinic visits. The physician/investigator will ask the patient if they have had any postoperative complications since their surgery and will be asked to detail any complications if they answer yes to this question. The investigators will also obtain permission to call the participants for a patient satisfaction questionnaire at 1 week post-op, and possibly 2 and 6 weeks if they have not presented for their post op/partum appointments or the questionnaire could not be obtained at their visit.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal Age 18 or above
2. Cesarean delivery
3. Maternal condition which increases the risk of wound complication. These conditions include: Obesity (BMI >30), diabetes, HIV/AIDS, chorioamnionitis, rheumatologic disease, history of wound complication, anticoagulant therapy.
4. Patient able to read and speak English or Spanish.

Exclusion Criteria:

1. Minors (<18 years of age)
2. Non-cesarean wound (ie tubal ligation wound)
3. No high risk maternal condition
4. Patient unable to read and speak English or Spanish.
5. Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Hill, MBBS, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez MG, Barske ME, Kjellsson KB, Saboda K, Reed HA, Hill MG. Topical negative pressure wound therapy to prevent wound complications following caesarean delivery in high-risk obstetric patients: A randomised controlled trial. Aust N Z J Obstet Gynaecol. 2023 Aug;63(4):516-520. doi: 10.1111/ajo.13675. Epub 2023 May 4. PMID 37140175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Dressing | PICO Dressing
Started | 75 | 79
Completed | 75 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing | PICO Dressing | Total
Number analyzed (Participants) | 75 | 79 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 79 | 154
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (6.5) | 30.5 (6.1) | 31.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 79 | 154
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 68 | 64 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United States | 75 | 79 | 154

OUTCOME MEASURES:

1. Primary Outcome: Wound Complication
Description: Number of study participants with a wound complication including wound breakdown, infection, separation or dehiscence
Time Frame: post operative day 1-42
Population: Participants who had any follow up at either 1, 2 or 6 weeks were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dressing | PICO Dressing
Number analyzed (Participants) | 67 | 71
Participants | 13 | 14

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Standard Dressing | PICO Dressing
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/79
Other Adverse Events (participants affected / at risk) | 0/75 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03082664/Prot_000.pdf